CLINICAL TRIAL: NCT04759521
Title: Evaluation of Liver Fibrosis in Chronic Hepatitis B Patients With 2D Shear Wave Elastography With Propagation Map: A Single Center Study
Brief Title: Evaluation of Liver Fibrosis With 2D-Shear Wave Elastography
Status: Completed | Type: Observational
Sponsor: Seyhmus Kavak (Other)
Responsible Party: Sponsor-Investigator, Seyhmus Kavak, MD, Radiologist, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Organization: Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other)
Other Study IDs: 2019/215
Record Dates: First submitted 2021-02-13; First posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Chronic Hepatitis B; Sonoelastography; Fibrosis, Liver
Keywords: Shear wave elastography; Propagation map; Chronic Hepatitis; Liver fibrosis
MeSH Terms: conditions — Hepatitis B, Chronic; Liver Cirrhosis; Hepatitis, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Inactive HBsAg carriers were patients with HBsAg positivity for more than 6 months
- Group 2: Patients diagnosed with chronic hepatitis B were patients with HBsAg positivity for more than 6 months
- Group 3: The control group was composed of healthy individuals who were not infected with hepatitis B virus and did not fit any exclusion criteria.

SUMMARY:
The aims of this study are to evaluate liver fibrosis with two-dimensional (2D) shear wave elastography (SWE) technique in inactive hepatitis B surface antigen (HBsAg) carriers and patients with active chronic hepatitis B (CHB), with the help of a propagation map, compare this method with histopathological results in patients with CHB and determine the suitability of 2D-SWE for use instead of liver biopsy by evaluating fibrosis before and after treatment.

DETAILED DESCRIPTION:
A total of 253 patients with CHB and inactive HBsAg carriers as well as a control group of 30 healthy individuals were included in the study between January 2019 and October 2020. Liver stiffness measurements with 2D-SWE, fibrosis-4 (FIB-4) and aspartate aminotransferase to platelet ratio index (APRI) scoring and additional liver biopsy in patients with CHB were performed in all cases with the help of the propagation map. Depending on the degree of fibrosis, liver stiffness was measured again at 24 and 48 weeks in patients who received antiviral therapy. Spearman rank correlation test was used for analysing correlation between variables, and receiver operating curve analysis was used to evaluate diagnostic performance in terms of fibrosis.

ELIGIBILITY:
Inclusion Criteria:

1. Being infected with the hepatitis B virus,
2. > 18 years old
3. < 64 years old

Exclusion Criteria:

1. Co-infection with hepatitis C or D
2. Have chronic or acute fulminant liver disease
3. Have DM disease
4. Hypertriglyceridemia, obesity, grade2 and higher hepatosteatosis,
5. Long-term drug use, alcohol intake that may damage the liver
6. Under the age of eighteen
7. Over sixty-five years old
8. Transplantation patients

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A total of 253 patients with CHB and inactive hepatitis B surface antigen (HBsAg) carriers who presented to the Infectious Diseases outpatient clinic were included in the study. In addition, a healthy control group of 30 people was included.
Sampling Method: Non-Probability Sample
Enrollment: 253 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
Comparison of liver stiffness levels of group 1 and group 2 patients | 1st week, 24th week and 48th week
  Liver stiffness levels of group 1 and group 2 patients were compared by measuring in kPa and m / s using 2D-SWE technique. Possible increase and decrease values in liver stiffness measurements were calculated at 24 and 48 weeks in subjects who received antiviral therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Sağlik Bilimleri Üniversitesi Training and Research Hospital, Diyarbakır, Turkey (Türkiye)